CLINICAL TRIAL: NCT01581489
Title: Early Versus Delayed Cord Clamping at Term: Neurodevelopmental Outcomes in Swedish Infants at 4 Years of Age
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Umeå University (Other); Halmstad County Hospital (Other); County Council of Halland, Sweden (Other Government)
Responsible Party: Sponsor
Other Study IDs: NATIBAR1213
Record Dates: First submitted 2012-03-13; First posted 2012-04-20 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Developmental Delay; Iron Deficiency
Keywords: Cord clamping; iron deficiency; Neurodevelopment
MeSH Terms: conditions — Learning Disabilities; Iron Deficiencies | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early cord clamping (ECC): Early cord clamping consisted of early (=< 10 s) clamping of the umbilical cord at birth.
  Interventions: Procedure: Time to clamping of the umbilical cord after delivery
- Delayed cord clamping (DCC): Delayed cord clamping consisted of delayed (>= 180 s) clamping of the umbilical cord at birth.
  Interventions: Procedure: Time to clamping of the umbilical cord after delivery

INTERVENTIONS:
Procedure: Time to clamping of the umbilical cord after delivery — The time after delivery of the newborn until the midwife stops the circulation in the umbilical cord with a clamp.
  Other Names: Immediate cord clamping; Late cord clamping; Deferred cord clamping

SUMMARY:
Delayed clamping of the umbilical cord might prevent or slow the onset of iron deficiency by increasing the infant's iron endowment at birth. Compared to early clamping, a delay in clamping in clamping of around 2-3 min provides an additional 25-40 mL of blood per kg of bodyweight to the newborn infant.

The results of previous intervention studies on delayed clamping are mixed, and few have followed the infants beyond the perinatal period. All longer follow up studies have been performed in low income countries except for the investigators earlier study, showing less iron deficiency and improved iron stores after delayed cord clamping at 4 months of age.

The main objective of the current study is to assess whether the time of cord clamping affects neurodevelopment at 4 years of age in a large sample of full-term, Swedish infants. The investigators hypothesis is that as delayed cord clamping improves iron stores at 4 months, this could affect the child's development positively.

DETAILED DESCRIPTION:
Project description

Iron deficiency is associated with neurodevelopmental delay and suboptimal cognitive function. Our hypothesis is that early cord clamping is associated with an increased risk for iron deficiency, and as a consequence increased risk for suboptimal infant development also in a country with high standard of living.

* Method

  1. Study cohort Four-hundred full-term infants, born to healthy mothers after normal pregnancies, were randomized to early or delayed cord clamping (at a hospital which practiced early cord clamping as standard practice). The infants were born during the time-period April 2008 to May 2009. Pregnant women were considered eligible if they met the following criteria: non-smoking, healthy mother (no haemolytic disease, no treatment with any of the following drugs: anticonvulsants, antidepressants, thyroid hormone, insulin, chemotherapy or cortisone), normal pregnancy (no preeclampsia, no diabetes, no prolonged rupture of membranes or signs of infection), single birth, term pregnancy (gestational age 37 +0 until 41 +6 weeks + days), expected vaginal delivery with cephalic presentation. Furthermore, the mother should be able to master Swedish well enough to understand the meaning of the study. Mothers were given written and oral information about the trial at the maternal health care centre from 34 weeks of gestational age. Mothers fulfilling the inclusion criteria at the time of admission to the delivery ward were again given written and oral information about the study by the attending midwife and written informed consent was obtained. Randomization was performed in advance by computer in blocks of 20. When delivery was imminent, the midwife opened a sealed envelope containing the treatment allocation. The intervention in the early cord clamping (ECC) group consisted of double clamping of the umbilical cord within 10 seconds of the infant's delivery, and arterial and venous blood sampling from the clamped segment within 10 min. The intervention in the delayed cord clamping (DCC) group consisted of late (≥ 180 s) clamping of the umbilical cord and arterial and venous blood sampling from the unclamped cord within 30 seconds after birth, while the midwife was holding the child below the level of the uterus. In both randomization groups, all children were initially kept about 20 cm below the level of the mother's uterus for 30 seconds and then placed on their mother's chest. All other aspects of obstetric care during labour and delivery were managed according to the standard practice of care at the study hospital. Oxytocin was administered to all mothers immediately after cord clamping. The final participating mother-infant pairs available for statistical analysis were 189 in the ECC group and 193 in the DCC group.
  2. Follow up at 4 years of age

     Children will be asked to return for a follow up at 4 years of age for neuro-developmental testing including:
     * Cognitive testing with WPPSI (Wechsler Preschool and Primary Scale of Intelligence)
     * Behavioral assessment with SDQ (Strengths and Difficulties Questionnaire), a questionnaire for behavioural screening which is filled in by the parents
     * Assessment of psychomotor development with ASQ (Ages and Stages Questionnaire), a questionnaire that is filled in by the parents
     * Selected items from Movement ABC (Assessment Battery for Children)

     Time plan The included children were born during the time period April 2008 to May 2009, and they will become 4 years during 2012 and 2013. We aim to test them at the age of 4 years (April 2012 to May 2013). Additional research ethics permission for the follow up has been approved. Permission to translate and use the Ages and Stages Questionnaire (ASQ) for scientific purposes, has been sought from the publisher Brooks Publishing (as already approved for the previous versions at 4, 12 and 36 months of age).
* Realization At approximately one month before the child's fourth birthday, the parents will receive a letter containing information about the study,including time and location for the testing, and the two questionnaires, SDQ and ASQ. The parents are asked to answer these questionnaires before the visit to the psychologist.

The parents has also been informed about the planned neurodevelopmental testing and questionnaires at 4 years of age when they had another scheduled visit when the child was three years of age. The parents have the opportunity to contact the research assistant who can change the time for the visit. After the neurodevelopmental testing, the parents will receive a written report, and if abnormal results are discovered, due action will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the earlier cord clamping trial
* Age between 48 and 51 months

Ages: 48 Months to 51 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The eligble population consists of a group of 382 children who were included in a trial (NCT01245296) and randomized to either early or delayed cord clamping. The parents will be asked for consent for their child to participate in the current follow up study.
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2012-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Intelligence quotient (IQ) as measured by the Wechsler Preschool and Primary Scale of Intelligence-III. | 48 months (plus 3 months)
  The Wechsler Preschool and Primary Scale of Intelligence (WPPSI) is an intelligence test designed for children ages 2 years 6 months to 7 years 3 months. A trained and experienced psychologist will perform the test and do the evaluation.

SECONDARY OUTCOMES:
Score of the different subsets of Wechsler Preschool and Primary Scale of Intelligence-III. | 48 months (plus 3 months)
  The subsets of the Wechsler Preschool and Primary Scale include Verbal and Performance IQ; the Processing Speed Quotient and a General Language Composite. Each subset will result in a score, the difference between the intervention groups will be assessed with an appropriate statistical method
Psychomotor development assessed by the Ages and Stages Questionnaire. | 48 months (plus 3 months)
  Ages and Stages Questionnaire is a parent report questionnaire available for developmental screening of children from one month to 5 ½ years. 30 questions are divided into 5 developmental domains (communication, gross motor, fine motor, problem solving and personal-social). Total score and scores within separate domains from the 48-month questionnaire will be assessed.
Fine motor skills assessed by the Movement Assessment Battery for Children-Second Edition. | 48 months (plus 3 months)
  The Performance Test of the the Movement Assessment Battery for Children contains 8 tasks. The tasks cover the following 3 areas: manual dexterity (3 items), ball skills (2 items), and static and dynamic balance (3 items). A psychologist will observe and record how the child performs the tasks.
Behaviour assessed by the Strengths and Difficulties Questionnaire or it's subscales. | 48 months (plus 3 months)
  All versions of the SDQ ask about 25 attributes, some positive and others negative. These 25 items are divided between 5 scales:emotional symptoms (5 items), conduct problems (5 items), hyperactivity/inattention (5 items) and peer relationship problems (5 items) added together to generate a total difficulties score (based on 20 items) and a separate scale concerning prosocial behavior (5 items).
Gender effect on the result of the developmental tests. | 48 months (plus 3 months)
  All results from WPPSI-III, ASQ, SDQ and Movement ABC will be statistically analysed to evaluate if the combination of gender and timing of cord clamping will affect the results.
Gestational age effect on the result of the developmental tests. | 48 months (plus 3 months)
  All results from WPPSI-III, ASQ, SDQ and Movement ABC will be statistically analysed to evaluate if the combination of gender and timing of cord clamping will affect the results.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Andersson, MD, Principal Investigator — Hospital of Halland, Halmstad; Barbro Lindquist, PhD, Principal Investigator — Hospital of Halland, Halmstad; Lena Hellström-Westas, Professor, Study Chair — Uppsala University
Locations (1):
- Hospital of Halland, Halmstad, Halmstad, Halland County, Sweden

REFERENCES:
- [Background] Andersson O, Hellstrom-Westas L, Andersson D, Domellof M. Effect of delayed versus early umbilical cord clamping on neonatal outcomes and iron status at 4 months: a randomised controlled trial. BMJ. 2011 Nov 15;343:d7157. doi: 10.1136/bmj.d7157. PMID 22089242
- [Result] Andersson O, Lindquist B, Lindgren M, Stjernqvist K, Domellof M, Hellstrom-Westas L. Effect of Delayed Cord Clamping on Neurodevelopment at 4 Years of Age: A Randomized Clinical Trial. JAMA Pediatr. 2015 Jul;169(7):631-8. doi: 10.1001/jamapediatrics.2015.0358. PMID 26010418